CLINICAL TRIAL: NCT04037358
Title: A Phase II Randomized Trial of RAdium-223 and SABR Versus SABR for oligomEtastatic Prostate caNcerS (RAVENS)
Brief Title: RAdium-223 and SABR Versus SABR for Oligometastatic Prostate Cancers
Acronym: RAVENS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J18147; IRB00188450 (Other: JHM IRB)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223

STUDY DESIGN:
Intervention Model Description: RAdium-223 and SABR Versus SABR (Stereotactic Ablative Radiotherapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radium-223 and SABR (Experimental): First radium-223 infusion will be within two weeks of SABR
  Interventions: Drug: Radium-223; Radiation: stereotactic ablative radiotherapy (SABR)
- SABR (Active Comparator): SABR(1-5 fractions) will be administered for all men
  Interventions: Radiation: stereotactic ablative radiotherapy (SABR)

INTERVENTIONS:
Drug: Radium-223 — Radium-223 plus SABR will be within two weeks.
  Arms: Radium-223 and SABR
Radiation: stereotactic ablative radiotherapy (SABR) — SABR 1-5 fractions

SUMMARY:
This is a Phase II non-blinded randomized study evaluating men with oligometastatic prostate cancer lesions randomized (1:1) to stereotactic ablative radiation therapy (SABR) versus SBAR + Radium-223. We are looking to determine the progression-free survival of men who have oligometastatic prostate cancer with at least one bone metastasis with stereotactic ablative radiation therapy (SABR) versus SABR + Radium-223.

DETAILED DESCRIPTION:
The metastatic capacity of prostate cancer (PCa) behaves along a spectrum of disease that contains an oligometastatic state where metastases are limited in number and location. The importance of local consolidation of all tumor deposits in oligometastatic disease to forestall further metastatic dissemination is now backed by small randomized studies. Our previous Baltimore ORIOLE randomized trial of stereotactic ablative radiation (SABR) alone, highly focused, high-dose radiation, versus observation in oligometastatic PCa final data demonstrate a progression-free survival (PFS) benefit of SABR alone. The patterns of failure from our ORIOLE trial in combination with prior data suggest one dominant mode of failure is from microscopic disease particularly those with bone-tropic biology. These are important early clinical data suggesting the existence of an oligometastatic state and the importance of local therapies in the management of these patients. Radiopharmaceutical therapy (RPT) approaches have not been applied in the oligometastatic space and thus the opportunity to target micrometastatic disease in conjunction with local consolidation of macroscopic disease with SABR has the potential to provide a curative paradigm for patients with oligometastatic PCa. We introduce the successor trial to ORIOLE called RAVENS that is a phase II randomized trial of SABR +/- the bone metastasis seeking RPT Xofigo in men with oligometastatic PCa. We hypothesize macroscopic prostate tumors support the growth of and help nurture future distant metastases and this process can be impacted most by total, macro- and microscopic, tumor consolidation. In addition, we hypothesize that circulating biomarkers can identify men with oligometastasis that benefit the most from SABR and RPT.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have at least one and up to three asymptomatic metastatic tumor(s) of the bone or soft tissue (with at least one bone metastasis) develop within the past 6-months that are ≤ 5.0 cm or <250 cm3
* Patient must have had their primary tumor treated with surgery and/or radiation.
* Histologic confirmation of malignancy (primary or metastatic tumor).
* PSADT <15 months. PSA doubling time (PSADT) will be calculated using as many PSA values that are available from time of relapse (PSA > 0.2). To calculate PSADT, the Memorial Sloan Kettering Cancer Center Prostate Cancer Prediction Tool will be used. It can be found at the following web site: https://www.mskcc.org/nomograms/prostate/psa-doubling-time.
* Patient may have had prior systemic therapy and/or ADT associated with treatment of their primary prostate cancer. Patient may have had ADT associated with salvage radiation therapy (to the primary prostate cancer or pelvis is allowed).
* PSA > 0.5 but <50.
* Testosterone > 125 ng/dL.
* Patient must be ≥ 18 years of age.
* Patient must have a life expectancy ≥ 12 months.
* Patient must have an ECOG performance status ≤ 2.
* Patient must have normal organ and marrow function as defined as:

Before the first administration of Xofigo, the absolute neutrophil count (ANC) should be ≥ 1.5 x 109/L, the platelet count ≥ 100 x 109/L and hemoglobin ≥ 10 g/dL.

* Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No more than 3 years of ADT is allowed, with the most recent ADT treatment having occurred greater than 6 months prior to enrollment.
* PSMA-PET/MRI or PSMA-PET/CT scan within the past 6 months with results that demonstrate more disease lesions than baseline CT/Bone Scan
* Castration-resistant prostate cancer (CRPC).
* Spinal cord compression or impending spinal cord compression.
* Suspected pulmonary and/or liver metastases (greater >10 mm in largest axis).
* Patient receiving any other investigational agents.
* Patient receiving abiraterone and prednisone.
* Patient is participating in a concurrent treatment protocol.
* Serum creatinine > 3 times the upper limit of normal.
* Total bilirubin > 3 times the upper limit of normal.
* Liver Transaminases > 5-times the upper limit of normal.
* Unable to lie flat during or tolerate PET/MRI, PET/CT or SBRT.
* Prior salvage treatment to the primary prostate cancer or pelvis is allowed.
* Refusal to sign informed consent.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kiess, M.D., Principal Investigator — Johns Hopkins SKCCC
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang JH, Sherry AD, Bazyar S, Sutera P, Radwan N, Phillips RM, Deek MP, Lu J, Dipasquale S, Deville C, DeWeese TL, Song DY, Wang H, Hobbs RF, Malek R, Dudley SA, Greco SC, Antonarakis ES, Marshall CH, Denmeade S, Paller CJ, Carducci MA, Pienta KJ, Oz OK, Ramotar M, Leenstra JL, Park SS, Abramowitz MC, Desai N, Berlin A, Stish BJ, Tang C, Tran PT, Kiess AP. Outcomes of Radium-223 and Stereotactic Ablative Radiotherapy Versus Stereotactic Ablative Radiotherapy for Oligometastatic Prostate Cancers: The RAVENS Phase II Randomized Trial. J Clin Oncol. 2025 Jun 20;43(18):2059-2068. doi: 10.1200/JCO-25-00131. Epub 2025 May 7. PMID 40334149
- [Derived] Hasan H, Deek MP, Phillips R, Hobbs RF, Malek R, Radwan N, Kiess AP, Dipasquale S, Huang J, Caldwell T, Leitzel J, Wendler D, Wang H, Thompson E, Powell J, Dudley S, Deville C, Greco SC, Song DY, DeWeese TL, Gorin MA, Rowe SP, Denmeade S, Markowski M, Antonarakis ES, Carducci MA, Eisenberger MA, Pomper MG, Pienta KJ, Paller CJ, Tran PT. A phase II randomized trial of RAdium-223 dichloride and SABR Versus SABR for oligomEtastatic prostate caNcerS (RAVENS). BMC Cancer. 2020 Jun 1;20(1):492. doi: 10.1186/s12885-020-07000-2. PMID 32487038

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radium-223 and SABR | SABR
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0
Not completed — Patient withdrew before intervention | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 and SABR | SABR | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Median (Full Range); unit: years] | 66 [55.0 to 86.0] | 69 [55 to 84] | 68 [55 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 33 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27 | 29 | 56
  African American | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Other | 1 | 0 | 1
  Hispanic/Latino | 2 | 2 | 4
  Not Hispanic/Latino | 28 | 31 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 28 | 53
  Canada | 5 | 5 | 10
International Society of Urological Pathology (ISUP) Group Grade [Count of Participants; unit: Participants] — ISUP grade group is a 5-tier system that categorizes the aggressiveness of prostate cancer. Grade Group 1 (lease aggressive) to Grade Group 5 (most aggressive). The ISUP group grade is based on corresponding Gleason scores.
  Grade group 1: (Gleason score <=6); Grade Group 2: (Gleason score 3+4 = 7); Grade Group 3: (Gleason score 4+3 = 7); Grade Group 4: (Gleason score 4+4 = 8. 3+5 = 8, or 5+3 = 8); Grade Group 5: (Gleason score 9 or 10)
  Participants
    ISUP Group Grade 1-3 | 17 | 12 | 29
    ISUP Group Grade 4-5 | 13 | 21 | 34
Initial Management/Treatment [Count of Participants; unit: Participants]
  Radiation | 5 | 7 | 12
  Surgery | 25 | 26 | 51
Previous Hormone Therapy [Count of Participants; unit: Participants]
  No | 9 | 11 | 20
  Yes | 21 | 22 | 43
Baseline PSA, ng/mL [Mean (Standard Deviation); unit: ng/mL] | 6.20 (8.24) | 5.08 (5.88) | 5.61 (7.06)
Initial Imaging Type [Count of Participants; unit: Participants]
  Conventional Only | 6 | 3 | 9
  Conventional and PSMA-PET | 9 | 8 | 17
  Conventional and non-PSMA-PET | 8 | 9 | 17
  PSMA -PET Only | 5 | 9 | 14
  Non-PSMA-PET Only | 2 | 4 | 6
Initial Lesion [Count of Participants; unit: Participants]
  Bone Only | 21 | 28 | 49
  Bone and Lymph node | 9 | 5 | 14
Total Lesion Number [Count of Participants; unit: Participants]
  1 Lesion | 14 | 20 | 34
  2 Lesions | 7 | 10 | 17
  3 Lesions | 8 | 2 | 10
  4 Lesions | 0 | 1 | 1
  5 Lesions | 1 | 0 | 1
Bone Lesions Number [Count of Participants; unit: Participants]
  1 | 20 | 24 | 44
  2 | 6 | 9 | 15
  3 | 4 | 0 | 4
Bone Lesions Type [Count of Participants; unit: Participants]
  No lesion outside pelvis/vertebra | 19 | 18 | 37
  Lesions outside pelvis/vertebra | 11 | 15 | 26
Extra-pelvic lymph nodes [Count of Participants; unit: Participants]
  No | 28 | 31 | 59
  Yes | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time to progression in men who have oligometastatic prostate cancer after therapy. Progression is defined by PCWG2 criteria as follows: >=25% increase in PSA from nadir (and by >=2ng/mL), and/or clinical/radiographic progression (clinical progression = symptomatic progression, worsening of disease-related symptoms or new cancer-related complications; radiographic progression on CT scan defined by RECIST 1.1 criteria: >=20% enlargement in sum diameter of soft-tissue target lesions; or on bone scan >=1 new bone lesions), initiation of ADT or death due to any cause, whichever occurs first.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 10.5 [7.30 to 12.40] | 11.8 [6.67 to 21.2]

2. Secondary Outcome: Toxicity as Assessed by Number of Participants Who Experience Adverse Events Grade 3 or Greater (CTCAE v4.0)
Description: Adverse events grade 3 or higher (defined by CTCAE v4.0) measured as treatment related events in either SABR or SABR and Radium-223 arms.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Participants
  Grade 3 or higher Adverse Events | 5 | 3
  Fatigue | 0 | 1
  Lymphocyte Count Decrease | 4 | 1
  Insomnia | 0 | 1
  Musculoskeletal Pain | 1 | 0

3. Secondary Outcome: Rate of Local Control at 12 Months
Description: Percentage of participants achieving local control at 12 months
Time Frame: Up to 12 months
Population: One patient in the SABR arm never received imaging (data not collected) afterward due to loss of follow up/died for other reasons, so that patient will be censored out or excluded.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 32
percentage of participants | 0.794 [0.628 to 1] | 0.908 [0.793 to 1]

4. Secondary Outcome: Time to Locoregional Progression
Description: Time from starting treatment until local and/or regional relapse is documented
Time Frame: 12 months
Population: There were no locoregional progression events at the site of SBRT during the time patients were on study.
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Distant Progression
Description: Time from starting treatment until distant relapse is documented
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 11.9 [8.6 to 15.1] | 12.1 [9.1 to NA] — Upper 95% confidence interval not able to be estimated. Not estimable as there were too few events at later time points.

6. Secondary Outcome: Metastasis-Free Survival
Description: Time from treatment start to the time of a newly documented tumor metastasis by CT and/or bone scan. Subjects who do not progress will be censored at the time of the last contact.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 12.3 [11.9 to NA] — Upper 95% confidence interval not able to be estimated. NA explanation is not estimable as there were too few events at later time points. | 19.4 [8.22 to NA] — Upper 95% confidence interval not able to be estimated. NA explanation is not estimable as there were too few events at later time points.

7. Secondary Outcome: Androgen-deprivation Therapy (ADT)-Free Survival
Description: Time from randomization until initiation of androgen-deprivation therapy (ADT). ADT Free Survival (ADT-FS) is defined as the time from starting treatment to the time of initiation of palliative ADT.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 16.2 [12.3 to NA] — Upper 95% confidence interval not able to be estimated. NA explanation is not estimable as there were too few events at later time points. Standard nomenclature. | 19.2 [12.0 to NA] — Upper 95% confidence interval not able to be estimated. NA explanation is not estimable as there were too few events at later time points.

8. Secondary Outcome: Quality of Life as Assessed by Pain Severity and Pain Interference Score With Imputations Using the Brief Pain Inventory
Description: The brief pain inventory assesses the severity of pain, location of pain, amount of pain over the last 24 hours, and impact of pain on daily functions. Scores for the 4 pain severity items and 7 pain interference items range from 0-10, where 10 is the worst pain or pain that completely interferes with described activity and 0 is the least pain or does not interfere with described activity. The mean of these scores is used to measure pain severity and pain interference.
Time Frame: Baseline, Day 360
Population: Participants with missing data, and further 2 participants were not assessed due to disease progression for SBRT group and SBRT+Ra223 group, respectively.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 28 | 30
score on a scale
  Baseline BPI Score | 0.31 [0.06 to 0.56] | 0.39 [0.01 to 0.77]
  Day 360 BPI Score: number analyzed (Participants) | 20 | 17
  Day 360 BPI Score | 0.56 [0.06 to 1.05] | 0.27 [-0.2 to 0.73]

9. Secondary Outcome: Change in Quality of Life as Assessed by Pain Severity and Pain Interference With Imputations Using the Brief Pain Inventory
Description: as for outcome 8
Time Frame: Baseline, Day 360
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 20 | 17
score on a scale | 0.34 [-0.07 to 0.74] | -0.01 [-0.13 to 0.11]

10. Secondary Outcome: Time to New Metastatsis
Description: Time to New Metastasis (TNM) is defined as the time from starting treatment to the time of a new documented tumor metastasis by CT and/or bone scan. Subjects who do not progress will be censored at the time of the last contact.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 11.9 [8.6 to 15.1] | 12.0 [8.2 to NA] — NA Explanation: Upper 95% confidence interval not able to be estimated. Not estimable as there were too few events at later time points.

11. Secondary Outcome: Duration of Response
Description: Response will be defined as evidence of CR, PR, or stable disease. The duration of response will be measured from the start of treatment until the criteria for progression are met
Time Frame: 12 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 and SABR | SABR
Number analyzed (Participants) | 30 | 33
Months | 10.5 [7.3 to 12.4] | 11.8 [6.7 to 21.2]

ADVERSE EVENTS:
Time Frame: From the time of enrollment to 1 year or until progression of disease (up to 2 years)
Description: CTCAE (4.0) Grade 3 or higher adverse events.
Arm/Group | Radium-223 and SABR | SABR
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 30/31 | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radium-223 and SABR (N=31) | SABR (N=33)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 16 | 6
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 13 | 7
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Lymphocute cound decreased (Investigations) | 23 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Weight loss (Investigations) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 — Decreased appetite
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 — Loose bowel Movements
Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Neutrophl count decreased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 9 | 0
Urinary Urgency (Renal and urinary disorders) | 1 | 0
Any Adverse Event (General disorders) | 27 | 21 — Number of patients whose worst AE was grade 1-2, 3 and total.

LIMITATIONS AND CAVEATS:
Treatment and follow-up occurred during the COVID-19 pandemic, leading to assessment biases associated with telemedicine encounters. This study was conducted before routine use of molecular imaging (not mandated) to corroborate disease burden detected on conventional imaging. The study size is small and limits the prognostic correlates observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT04037358/Prot_SAP_000.pdf